CLINICAL TRIAL: NCT07162961
Title: A Single-center, Randomized, Prospective, Controlled Clinical Study on the Efficacy of Nintedanib in Improving Reproductive Outcomes in Women With Adenomyosis
Brief Title: Nintedanib for Improving Reproductive Outcomes in Adenomyosis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Assistant Dean, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: New IVF
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Adenomyosis of Uterus
Keywords: Adenomyosis; nintedanib
MeSH Terms: conditions — Adenomyosis | interventions — nintedanib; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nintedanib + Progesterone (Experimental): Nintedanib Esylate Soft Capsules (100mg). Oral, twice daily (BID) for 3 months+ Progesterone therapy (as per standard practice for 3 months).
  Interventions: Drug: Nintedanib; Drug: Progesterone
- Progesterone Only (Active Comparator): Progesterone therapy (as per standard practice for 3 months).
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Nintedanib — Participants will be randomly assigned to one of two groups: the Experimental Group will receive oral nintedanib (100 mg twice daily) plus progesterone therapy for three months; the Control Group will receive progesterone therapy only.
  Arms: Nintedanib + Progesterone
Drug: Progesterone — For control group

SUMMARY:
This study aims to evaluate the effectiveness and safety of nintedanib, an antifibrotic drug, in improving live birth rates for infertile women with adenomyosis who have frozen embryos. Based on promising animal data showing reduced uterine fibrosis, participants will be randomized to receive either standard progesterone therapy plus nintedanib or progesterone therapy alone for three months before undergoing a frozen embryo transfer cycle.

ELIGIBILITY:
Inclusion Criteria:

Aged 20-38, diagnosed with primary or secondary infertility; with at least one vitrified high-quality blastocyst (grading ≥4BB).

Diagnosed with adenomyosis within the last 3 months by MRI or transvaginal ultrasound, meeting the criteria of the Chinese Expert Consensus on Diagnosis and Treatment of Adenomyosis.

Body Mass Index (BMI) between 18-27 kg/m².

Regular menstrual cycles, no amenorrhea or severe dysfunctional uterine bleeding.

Normal ovarian reserve (AMH > 1 ng/mL or AFC ≥ 5 per ovary), not currently receiving ovarian suppression therapy.

Signed informed consent, able to understand and voluntarily participate, and willing not to participate in other clinical trials during the study period.

Exclusion Criteria:

Uterine or adnexal abnormalities (e.g., intrauterine adhesions, unicornuate/bicornuate/arcuate uterus, unremoved hydrosalpinx, endometrial polyp, submucosal myoma, or intramural myoma distorting the endometrial cavity).

History of GnRH agonist injection within 3 months prior to embryo transfer.

Unexplained abnormal vaginal bleeding.

Known active pelvic inflammatory disease.

Known genital malformation unsuitable for pregnancy.

Abnormal cervical cytology (TCT) results within 1 year before screening.

Severe impairment of liver or kidney function, heart disease, or hypertension.

Known history of thrombophlebitis or thromboembolic disease.

Any known clinically significant systemic disease (e.g., diabetes, tuberculosis).

Known history of recurrent miscarriage.

Chromosomal karyotype abnormality in either partner.

Either partner has a genetic disease deemed unsuitable for childbearing per the "Maternal and Infant Health Care Law".

Either partner has been exposed to teratogenic levels of radiation, toxins, or drugs.

Any condition/combined surgery/medication/other clinically significant abnormal lab finding judged by the investigator to potentially affect trial results.

Known refusal or inability to comply with the protocol requirements for any reason.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 328 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
live birth rate | Up to approximately 9-12 months after embryo transfer (considering gestation)
  Defined as the delivery of any live infant after 24 weeks of gestation. Calculated as: (Number of subjects with live birth / Number of subjects undergoing embryo transfer) * 100%.

IPD SHARING:
Plan to Share IPD: No
This involves the patient's informed consent.